CLINICAL TRIAL: NCT02239289
Title: Correction of Abnormal Flexion-relaxation Phenomenon in Chronic Low Back Pain: the Benefit Associated With Biofeedback Training
Brief Title: Use of Biofeedback Training to Correct Abnormal Neuromechanical Pattern in Chronic Low Back Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec à Trois-Rivières (Other)
Responsible Party: Principal Investigator, Martin Descarreaux, Professor, Université du Québec à Trois-Rivières
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIR UQTR 2013-2014
Record Dates: First submitted 2014-09-04; First posted 2014-09-12 (Estimated); Results first posted 2015-07-23 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Chronic Low Back Pain; Mechanical Low Back Pain
Keywords: Low back pain; Rehabilitation; Biofeedback; Electromyography; Kinematic
MeSH Terms: conditions — Low Back Pain | interventions — Biofeedback, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Biofeedback (Experimental): Subjects will be provided with four sessions of supervised biofeedback training
  Interventions: Other: Biofeedback

INTERVENTIONS:
Other: Biofeedback — Idem as described in the arm section (above)

SUMMARY:
The purpose of the present study is to evaluate the benefit of biofeedback training on the capacity of chronic low back pain patients to decrease their lumbar paraspinal muscles activity during trunk full flexion and its relationship with changes in clinical outcomes. To do so, twenty patients with nonspecific mechanical low back pain will be recruited and all participants will take part in four sessions of supervised biofeedback training, consisting of 5 blocks with at least 12 trunk flexion-extension tasks. It is hypothesized that participants will have improved neuromechanical parameters with the biofeedback training and that this improvement will be positively associated to changes in clinical outcomes. This study will also allow for generation of preliminary data, in order to plan for a larger randomized control trial.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18 and 60 years of age.
* Presence of non-specific chronic low back pain.

Exclusion Criteria:

* Prior surgery or major spine trauma.
* Lumbar scoliosis greater than 20°.
* Neuromuscular disease.
* Malignant tumor.
* Uncontrolled hypertension.
* Infection.
* Neurological deficit.
* Symptomatic lumbar disc herniation.
* Pregnancy.
* Recent lumbar cortisone injection.
* Active lower body injury and/or disabling pain limiting the capacity to complete the experimentation.
* Being under medications known to impair physical effort and pain perception.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2014-03; Primary Completion 2014-09 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Descarreaux, DC, PhD, Principal Investigator — Université du Québec à Trois-Rivières
Locations (1):
- Université du Québec à Trois-Rivières, Trois-Rivières, Quebec, Canada

REFERENCES:
- [Background] Giggins OM, Persson UM, Caulfield B. Biofeedback in rehabilitation. J Neuroeng Rehabil. 2013 Jun 18;10:60. doi: 10.1186/1743-0003-10-60. PMID 23777436
- [Background] Frank DL, Khorshid L, Kiffer JF, Moravec CS, McKee MG. Biofeedback in medicine: who, when, why and how? Ment Health Fam Med. 2010 Jun;7(2):85-91. PMID 22477926
- [Background] Hodges PW. Pain and motor control: From the laboratory to rehabilitation. J Electromyogr Kinesiol. 2011 Apr;21(2):220-8. doi: 10.1016/j.jelekin.2011.01.002. PMID 21306915
- [Background] Demoulin C, Crielaard JM, Vanderthommen M. Spinal muscle evaluation in healthy individuals and low-back-pain patients: a literature review. Joint Bone Spine. 2007 Jan;74(1):9-13. doi: 10.1016/j.jbspin.2006.02.013. Epub 2006 Nov 13. PMID 17174584

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Biofeedback
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Biofeedback
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.52 (11.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 13
Region of Enrollment [Number; unit: participants]
  Canada | 21
Body mass index, mean (SD) [Mean (Standard Deviation); unit: kg/m^2] | 22.55 (3.86)
Duration of low back pain in months, mean (SD) [Mean (Standard Deviation); unit: months] | 88.36 (65.26)
Fear of movement level [Mean (Full Range); unit: Units on a scale] — Tampa scale for kinesiophobia ranges from 1 to 68. Higher score indicates a higher fear of movement level.
  Units on a scale | 32.76 [22 to 48]
Disability level [Mean (Full Range); unit: units on a scale] — Oswestry disability index ranges from 0 to 100. Higher score indicates a higher lumbar disability level.
  units on a scale | 12.95 [0 to 28]
Current pain intensity [Mean (Full Range); unit: Units on a scale] — 101-points numerical rating scale that ranges from 0 (no pain) to 100 (worst possible pain).
  Units on a scale | 18.24 [0 to 65]
Pain intensity in the past week [Mean (Full Range); unit: Units on a scale] — 101-points numerical rating scale that ranges from 0 (no pain) to 100 (worst possible pain).
  Units on a scale | 24.62 [0 to 60]

OUTCOME MEASURES:

1. Primary Outcome: Flexion-relaxation Ratio
Description: Flexion-relaxation ratio is calculated by dividing muscle activity (EMG) during trunk flexion by muscle activity during full-flexed position. EMG of lumbar paraspinal muscles is recorder through surface EMG during every trials of each session.
Time Frame: Week 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Biofeedback
Number analyzed (Participants) | 21
Ratio | 0.68 (0.24)

2. Primary Outcome: Flexion-relaxation Ratio
Description: as for outcome 1
Time Frame: Week 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Biofeedback
Number analyzed (Participants) | 21
ratio | 0.76 (0.18)

3. Primary Outcome: Flexion-relaxation Ratio
Description: as for outcome 1
Time Frame: Week 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Biofeedback
Number analyzed (Participants) | 21
ratio | 0.76 (0.16)

4. Primary Outcome: Flexion-relaxation Ratio
Description: as for outcome 1
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Biofeedback
Number analyzed (Participants) | 21
ratio | 0.75 (0.18)

5. Secondary Outcome: Lumbo-pelvic Range of Motion During Trunk Flexion-extension
Description: Range of motion is recorder throught 8 kinematic markers placed on the right lower limb and the back of each participant during every trials of each session.
Time Frame: Week 1
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Biofeedback
Number analyzed (Participants) | 21
Degrees
  Pelvic range | 44.03 (9.13)
  Lumbar range | 45.15 (9.66)

6. Secondary Outcome: Disability Level
Description: Oswestry disability index ranges from 0 to 100. A higher score indicates higher disability.
Time Frame: Week 4
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Biofeedback
Number analyzed (Participants) | 21
units on a scale | 14.70 [0 to 44]

7. Secondary Outcome: Pain Intensity in the Past Week
Description: 101-points numerical rating scale that ranges from 0 (no pain) to 100 (worst possible pain).
Time Frame: Week 2
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Biofeedback
Number analyzed (Participants) | 21
Units on a scale | 22.90 [10 to 60]

8. Secondary Outcome: Current Pain Intensity
Description: 101-points numerical rating scale that ranges from 0 (no pain) to 100 (worst possible pain).
Time Frame: Week 3
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Biofeedback
Number analyzed (Participants) | 21
Units on a scale | 22.62 [0 to 80]

9. Secondary Outcome: Fear of Movement Level
Description: Tampa scale for kinesiophobia ranges from 0 to 68. Higher score indicates higher fear of movement level.
Time Frame: Week 4
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Biofeedback
Number analyzed (Participants) | 21
units on a scale | 29.80 [0 to 49]

10. Secondary Outcome: Current Pain Intensity
Description: 101-points numerical rating scale that ranges from 0 (no pain) to 100 (worst possible pain).
Time Frame: Week 2
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Biofeedback
Number analyzed (Participants) | 21
Units on a scale | 17.19 [0 to 50]

11. Secondary Outcome: Current Pain Intensity
Description: 101-points numerical rating scale that ranges from 0 (no pain) to 100 (worst possible pain).
Time Frame: Week 4
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Biofeedback
Number analyzed (Participants) | 21
Units on a scale | 19.81 [0 to 80]

12. Secondary Outcome: Pain Intensity in the Past Week
Description: 101-points numerical rating scale that ranges from 0 (no pain) to 100 (worst possible pain).
Time Frame: Week 3
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Biofeedback
Number analyzed (Participants) | 21
Units on a scale | 21.48 [0 to 80]

13. Secondary Outcome: Pain Intensity in the Past Week
Description: 101-points numerical rating scale that ranges from 0 (no pain) to 100 (worst possible pain).
Time Frame: Week 4
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Biofeedback
Number analyzed (Participants) | 21
Units on a scale | 23.62 [5 to 80]

14. Secondary Outcome: Lumbo-pelvic Range of Motion During Trunk Flexion-extension
Description: as for outcome 5
Time Frame: Week 2
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Biofeedback
Number analyzed (Participants) | 21
Degrees
  Pelvic range | 44.45 (8.26)
  Lumbar range | 48.60 (11.64)

15. Secondary Outcome: Lumbo-pelvic Range of Motion During Trunk Flexion-extension
Description: as for outcome 5
Time Frame: Week 3
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Biofeedback
Number analyzed (Participants) | 21
Degrees
  Pelvic range | 47.38 (9.15)
  Lumbar range | 47.83 (10.42)

16. Secondary Outcome: Lumbo-pelvic Range of Motion During Trunk Flexion-extension
Description: as for outcome 5
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Biofeedback
Number analyzed (Participants) | 21
Degrees
  Pelvic range | 47.21 (9.43)
  Lumbar range | 47.89 (9.16)

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: Only pain intensity was collected for adverse events by asking participants if their pain intensity increased at each session beginning.
Arm/Group | Biofeedback
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No